CLINICAL TRIAL: NCT07317492
Title: Prospective Evaluation of the Association Between Hemorrhoids and Lower Extremity Varicose Veins Using Doppler Ultrasound (HEMOVAR Study)
Brief Title: HEMOVAR Study on Hemorrhoids and Varicose Veins
Acronym: HEMOVAR
Status: Recruiting | Type: Observational
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Akay Edizsoy, Assistant Professor of General Surgery, Aydin Adnan Menderes University
Other Study IDs: HEMOVAR-ADU-2025-01; 2025/299-24 (Other: Aydın Adnan Menderes University Faculty of Medicine Local Ethics Committee Approval Number)
Record Dates: First submitted 2025-12-16; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Varicose Veins of Lower Limb; Hemorrhoids
Keywords: Hemorrhoids; Varicose Veins; Venous Insufficiency; Doppler Ultrasound; Venous Reflux; Proctology; Pelvic Congestion Syndrome; Prospective Observational Study; Varicocele; HEMOVAR Study
MeSH Terms: conditions — Hemorrhoids; Varicose Veins; Venous Insufficiency; Varicocele

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hemorrhoid Group: Adult patients (≥18 years) diagnosed with hemorrhoidal disease presenting to the general surgery proctology clinic.
- Control Group: Adult patients (≥18 years) with non-hemorrhoidal benign proctologic diseases presenting to the same clinic.

SUMMARY:
The HEMOVAR Study is a prospective observational study designed to evaluate the association between hemorrhoidal disease and lower extremity varicose veins. A total of 400 adult patients presenting to the general surgery proctology outpatient clinic of Aydın Adnan Menderes University Hospital will be included. The study will consist of two groups: 200 patients diagnosed with hemorrhoids and 200 patients with other non-hemorrhoidal benign proctologic conditions serving as controls.

All participants will undergo routine clinical evaluation and demographic data collection. Cardiovascular surgeons will voluntarily perform physical examination and Doppler ultrasonography of the lower extremities to assess venous insufficiency and varicose veins. No experimental intervention or treatment will be applied. The study will not require any consumable materials and will not impose any additional financial burden on the hospital, patients, or the national health insurance system. The primary outcome is the prevalence of lower extremity venous insufficiency in patients with hemorrhoids compared with controls.

DETAILED DESCRIPTION:
The HEMOVAR Study is a single-center, prospective, cross-sectional observational investigation conducted at Aydın Adnan Menderes University Hospital. The study aims to examine the association between hemorrhoidal disease and lower extremity venous insufficiency using standardized clinical assessment and Doppler ultrasonography. Adult patients presenting to the general surgery proctology outpatient clinic will be screened for eligibility and enrolled after providing written informed consent.

Two parallel groups will be formed: patients with clinically diagnosed hemorrhoids and a control group consisting of patients with other benign non-hemorrhoidal proctologic conditions. Cardiovascular surgeons will voluntarily perform clinical examination and color Doppler ultrasonography of the lower limb venous system in all participants. Doppler parameters including the presence of venous reflux, affected venous segments, reflux duration, venous diameter, and CEAP clinical classification will be recorded. Laboratory evaluation will be limited to hemoglobin measurement. Secondary analyses will explore the coexistence of other venous disorders such as varicocele and pelvic congestion syndrome.

This study involves no experimental intervention, randomization, or invasive procedures. No consumables will be used, and there will be no additional financial burden on the hospital, patients, or the national health insurance system. The study will commence following approval by the local ethics committee, and data will be collected and analyzed in accordance with the Declaration of Helsinki and Good Clinical Practice principles.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Patients presenting to the general surgery proctology outpatient clinic of Aydın Adnan Menderes University Hospital
* Patients diagnosed with hemorrhoidal disease or other non-hemorrhoidal benign proctologic conditions
* Ability to understand the study procedures and provide written informed consent

Exclusion Criteria:

* Patients younger than 18 years
* History of lower extremity varicose vein surgery, endovenous ablation, or sclerotherapy
* Presence of systemic venous disorders such as portal hypertension or liver cirrhosis
* Pregnant women
* Patients with known malignancy or severe comorbid conditions that could interfere with evaluation
* Refusal or inability to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients presenting to the general surgery proctology outpatient clinic with hemorrhoidal disease or other benign non-hemorrhoidal proctologic conditions.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-12-19 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Correlation between Hemorrhoidal Disease and Lower Extremity Venous Insufficiency | Baseline (single visit)
  The correlation between the presence of hemorrhoidal disease (yes/no) and lower extremity venous insufficiency will be assessed using color Doppler ultrasonography. Venous insufficiency will be defined as the presence of venous reflux lasting ≥0.5 seconds in superficial veins or ≥1.0 second in deep veins. The outcome will be expressed as the percentage of patients with Doppler-confirmed venous insufficiency in each study group.

SECONDARY OUTCOMES:
Correlation between Hemorrhoid Grade and Severity of Venous Insufficiency | Baseline (single visit)
  The correlation between hemorrhoid grade (Grade I-IV, assessed by clinical examination) and the severity of lower extremity venous insufficiency will be evaluated. Venous severity will be assessed using the CEAP clinical classification determined by Doppler ultrasonography. The outcome will be analyzed using correlation coefficients between hemorrhoid grade and CEAP class.

CONTACTS AND LOCATIONS:
Overall Officials: Akay Edizsoy, Assist Prof., Study Chair — Aydin Adnan Menderes University, School of Medicine
Locations (1):
- Aydin Adnan Menderes University Hospital, Aydin, Efeler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared outside of anonymized aggregate analyses.

REFERENCES:
- [Background] Salnikova LE, Khadzhieva MB, Kolobkov DS. Biological findings from the PheWAS catalog: focus on connective tissue-related disorders (pelvic floor dysfunction, abdominal hernia, varicose veins and hemorrhoids). Hum Genet. 2016 Jul;135(7):779-95. doi: 10.1007/s00439-016-1672-8. Epub 2016 Apr 28. PMID 27126235
- [Background] Ekici U, Kartal A, Ferhatoglu MF. Association Between Hemorrhoids and Lower Extremity Chronic Venous Insufficiency. Cureus. 2019 Apr 19;11(4):e4502. doi: 10.7759/cureus.4502. PMID 31249764
- [Background] Holdstock JM, Dos Santos SJ, Harrison CC, Price BA, Whiteley MS. Haemorrhoids are associated with internal iliac vein reflux in up to one-third of women presenting with varicose veins associated with pelvic vein reflux. Phlebology. 2015 Mar;30(2):133-9. doi: 10.1177/0268355514531952. Epub 2014 Apr 22. PMID 24755923